CLINICAL TRIAL: NCT02226679
Title: An Open Label Rollover Trial for Patients Randomized to the Control Group of Study LSH-10-001 (Rollover Study for AUGMENT-HF)
Brief Title: An Open Label Rollover Trial for Patients Randomized to the Control Group of Study LSH-10-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LoneStar Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSH-11-001
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure; Cardiomyopathy; Dilated Cardiomyopathy
Keywords: crossover; rollover study; open label
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Algisyl-LVR device implantation (Experimental): Algisyl-LVR™ employed as a method of left ventricular augmentation and restoration in patients with dilated cardiomyopathy. Algisyl-LVR™ will be injected into the myocardium under direct visualization during the surgical procedure.
  Interventions: Device: Algisyl-LVR

INTERVENTIONS:
Device: Algisyl-LVR — Algisyl-LVR™ device (implants) administered during a surgical procedure

SUMMARY:
The objective of this extension study is to evaluate the safety and potential beneficial effects of the Algisyl-LVR™ device in patients with established heart failure secondary to a dilated cardiomyopathy. The results of this study will provide confirmatory evidence of the long-term safety and effectiveness of the Algisyl-LVR in patients with established heart failure.

DETAILED DESCRIPTION:
This is a prospective, open-label evaluation of the safety and effectiveness of Algisyl-LVR in patients with dilated cardiomyopathy of either ischemic or non-ischemic origin. The evaluation for the primary measure of efficacy (Peak VO2) at 6 months will be investigator-blinded. The primary safety endpoint, while not blinded, is 30 day all-cause mortality and an objective assessment. The remaining study endpoints will evaluate the effects of the device through the evaluation of functional, structural, biochemical, and electrocardiographic evaluations at 6 and 12 months. Evaluation of adverse events and these assessments will also provide evidence of the safety profile of the device in patients with dilated cardiomyopathy.

Pre-enrollment baseline patient evaluation will include clinical assessment, assessment of New York Heart Association (NYHA) functional class, blood tests, transthoracic echocardiography, MRI, electrocardiogram, cardiopulmonary exercise testing (CPX), submaximal exercise testing, and quality of life assessments. Blinded central evaluation will be performed for measures of cardiopulmonary exercise testing and cardiac imaging.

*Note: The local CPX and echocardiography measurements will be used to determine patient eligibility with respect to the peak V02 values, ejection fraction and the left ventricular end diastolic dimension indexed to body surface area (LVEDDi). The core lab values for these same assessments will be used in all statistical analyses of the study.

Patient's eligible for this study completed at least 12 months of follow in the control group of the lead-in study LSH-10-001 and provided a written informed consent to participate in study LSH-001. A written informed consent to be enrolled in study LSH-11-001 is required for all patients electing participation in this roll-over study. After written patient informed consent has been obtained and verification of eligibility, patients who meet the inclusion and exclusion criteria can be included in the study and will have the Algisyl-LVR™ device (implants) administered during a surgical procedure. Patients will be considered part of this study cohort as soon as they have been hospitalized to receive the Algisyl-LVR device. The investigator will complete the "Premature Withdrawal from Follow-up" form in the patient's eCRF for study LSH-10-001 and indicate "Patient will receive the Algisyl-LVR device" as the reason for premature withdrawal from LSH-10-001. The acute response to device implant will be monitored intraoperatively via continuous electrocardiographic cardiac monitoring, arterial pressure lines, transesophageal echocardiography (TEE), and pulmonary artery catheter. Patients receiving the investigational device are expected to remain hospitalized for 5 to 14 days.

Follow-up in this study is divided into two phases. During the first phase, referred to as the "efficacy phase", repeat testing of patient functional and cardiac structural parameters will be conducted at follow-up visits scheduled at 3 months and 6 months, and every 6 months thereafter. Follow-up testing will be supplemented by a 30 day (post implant) telephone contact with all patients. The efficacy phase of the trial will end on a common closing date after a minimum of 6 months of follow-up (i.e., after the last patient enrolled has been completed the 6 month visit). At that point data analysis will be performed and an initial study report will be generated. Following completion of the efficacy phase, long-term monitoring will continue through each patient's 24-month visit. This second phase is referred to as the "extended follow-up phase". During this phase, data collection will be focused on long-term safety and will be conducted at 6-month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed at least 12 months of follow in the control group of the lead-in study LSH-10-001 are eligible to participate.

   Patients must have completed all study related procedures for the 12 month, 18 month or 24 month visit in Protocol LSH-10-001. Study procedures completed for the 12, 18 or 24 month visit in study LSH1-10-001 will be used as the baseline (screening) and qualifying procedures for study LSH-11-001 if the procedure was performed within 60 days of the date of Algisyl-LVR implant (screening procedures outside this window must be repeated).
2. The patients must be able and willing to give written informed consent
3. The patients will be adult (age ≥ 18 years and ≤ 79 years) males or females
4. The patients must be on stable, evidence-based therapy for heart failure

   Evidence-based therapy for heart failure is defined as an ACE-inhibitor (ACE-I), and/or angiotensin II receptor blockers (ARB) for patients at stable doses for 1 month prior to enrollment, if tolerated, and a beta blocker (carvedilol, metoprolol succinate, Nebivolol or bisoprolol) for 3 months prior to enrollment, if tolerated. Recent up-titration of the beta blocker is acceptable if the patient has been stable on this dose for 1 month prior to enrollment. Stable is defined as no more than a 100% increase or a 50% decrease in dose. Contraindications or intolerance to therapies should be documented. In those intolerant to both ACE-I and ARB, combination therapy with hydralazine and oral nitrate should be considered. Therapeutic equivalence for ACE-I substitutions is allowed within the enrollment stability timelines. Aldosterone inhibitor therapy should be added when NYHA Class III or IV symptoms occur on standard therapy. If aldosterone inhibitor therapy is to be administered in NYHA Class II patients, it must be initiated and optimized prior to enrollment. Eplerenone requires dosage stability for 1 month prior to enrollment. Diuretics should be used as necessary to keep the patient euvolemic. All heart failure therapeutics and dosages should be documented in the Case Report Forms.

   * Note: CRT or CRT-D are acceptable co-therapy, if placed > 3 months before implant of Algisyl-LVR or the investigator does not anticipate within 6 months after enrollment
5. The patients will have a left ventricular ejection fraction equal to or less than 35% via echocardiography, cardiac catheterization, radionuclide scan, or magnetic resonance imaging (measured within the last 30 days)
6. The patients will have a left ventricular end diastolic dimension indexed to body surface area (LVEDDi) of 30 to 40mm/m2 (LVEDD/BSA) (measured within the last 30 days).
7. Patients must have symptomatic heart failure with a Peak VO2 of 9.0 - 14.5 ml/min/kg (performed using a bicycle ergometer). Patients must perform two CPX tests (within 60 days of the Algisyl-LVR procedure and performed at least 20 hours apart) that differ by no more than 15% in the observed value for Peak VO2 and have a mean value of 9.0 - 14.5 ml/min/kg from these two tests.
8. Patient's surgical risk must be considered reasonable and the evaluation of surgical risk should include review of coronary and left ventricular angiography.
9. If female, the patients must be (a) post-menopausal, (b) surgically sterile, or (c) using adequate birth control and have a negative serum pregnancy test within 7 days prior to administration of study device.

Exclusion Criteria:

1. Patients for whom it is planned to receive CABG, MVR, heart transplantation or LVAD within the next 6 months
2. Patients presenting with cardiogenic shock
3. Patients who have undergone a previous mid-sternotomy surgical procedure are excluded unless the surgeon's assessment is that the left sided limited thoracotomy is feasible and considered reasonable surgical risk
4. Patients presenting with a restrictive cardiomyopathy such as due to amyloidosis, sarcoidosis, or hemochromatosis
5. Patient with a history of constrictive pericarditis
6. Patients with a Q wave myocardial infarction (MI) within the last 30 days
7. Patients with a recent history of stroke (within 60 days prior to the surgical procedure)
8. A left ventricular (LV) wall thickness of the LV free-wall, at the mid-ventricular level, of less than 8 mm (screening echocardiography must confirm a minimum wall thickness of 8 mm)
9. Patients with a serum creatinine > 2.5 mg/dL
10. Clinically significant liver enzyme abnormalities, i.e., AST(SGOT) and ALT (SGPT) more than 2.5 times the upper limit of normal
11. History of severe COPD (i.e., FEV 1< 1 liter or FEV1 < 50% predicted)
12. The patients will not be receiving concurrently an investigational Product in another clinical trial or have received an investigational Product in another clinical trial in the 30 days prior to enrollment
13. A life expectancy of less than 1 year or any other condition that, in the opinion of the clinical investigator, might compromise any aspect of the trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
estimate the 30 day mortality associated with the implantation of the Algisyl-LVR device | 30 days
  The primary safety objective is to estimate the 30 day mortality associated with the implantation of the Algisyl-LVR device

OTHER OUTCOMES:
Change in Peak VO2 from baseline to 6 months of follow-up | 6 months
  Change in Peak VO2 from baseline to 6 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ionel Droc, MD, Principal Investigator — Emergency Clinic Center for The Army For the Cardiovascular Diseases
Locations (2):
- A.O. Istituti Ospitalieri di Cremona"., Cremona, Italy
- Emergency Clinic Center of The Army for The Cardiovascular Diseases, Bucharest, Romania